CLINICAL TRIAL: NCT03610399
Title: Efficacy of Three Regimens of Chloroquine and Primaquine for the Treatment of Plasmodium Vivax Malaria in Cruzeiro do Sul, Acre, Brazil
Brief Title: Efficacy of 3 Regimens of Chloroquine and Primaquine for Treatment of P. Vivax Malaria, Cruzeiro do Sul, Acre, Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Brazil (Other Government); Evandro Chagas National Institute of Infectious Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7061
Record Dates: First submitted 2018-02-12; First posted 2018-08-01 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-06

CONDITIONS: P Vivax; Malaria, Vivax
Keywords: treatment response; efficacy; primaquine; chloroquine
MeSH Terms: conditions — Malaria, Vivax | interventions — Primaquine

STUDY DESIGN:
Intervention Model Description: We plan to compare 3 different regimens of primaquine for P. vivax treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Primaquine Regular Dose Unsupervised (Other): This is the regular primaquine dose Brazil without directly observed therapy.
  Interventions: Drug: Primaquine
- Primaquine Regular Dose Supervised (Active Comparator): This is the regular primaquine dose in Brazil but with directly observed therapy.
  Interventions: Drug: Primaquine
- Primaquine Double Dose Unsupervised (Active Comparator): This is the double total primaquine dose (14 days) in Brazil with directly observed therapy.
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — Different total dose and supervision.
  Other Names: Primaquine dose

SUMMARY:
We plan to assess the efficacy of 3 different regimens of chloroquine and primaquine for the treatment of P. vivax infections in Cruzeiro do Sul, Acre, Brazil. Patients will be divided in 3 different groups: treatment with regular dose of primaquine (0.5 mg/kg per day for 7 days) with directly observed therapy; regular dose of primaquine without directly observed therapy; and increased total dose of primaquine (0.5 mg/kg per day for14 days) with directly observed therapy. All patients will receive chloroquine (CQ) for three days at a daily dose of approximately 25 mg/Kg in accordance with the Brazilian National Malaria Control guidelines. Clinical and parasitologic parameters will be monitored over a 28-day follow-up period to evaluate drug efficacy and for a total period of 168 days (24 weeks) to evaluate chances of recrudescence, relapse, or reinfection. Results from this drug efficacy study will be used to assist the Brazilian Ministry of Health in assessing their national malaria treatment policy for P. vivax malaria.

DETAILED DESCRIPTION:
Background: The World Health Organization recommends that antimalarial treatment policies be evaluated every few years to check their efficacy. P. vivax malaria is the most common species in Brazil and cases are concentrated in the Amazon Region in Brazil.

Objectives: Assess the efficacy of 3 different regimens of chloroquine and primaquine for the treatment of P. vivax infections in Cruzeiro do Sul, Acre, Brazil.

Methods: An in vivo drug efficacy study will be conducted in Cruzeiro do Sul, Acre State, Brazil. A total of 257 study participants ≥5 years of age with parasitologically confirmed P. vivax monoinfections will be included. Patients will be divided in 3 different groups: treatment with regular dose of primaquine (0.5 mg/kg per day for 7 days) with directly observed therapy; regular dose of primaquine without directly observed therapy; and increased total dose of primaquine (0.5 mg/kg per day for14 days) with directly observed therapy. All patients will receive chloroquine (CQ) for three days at a daily dose of approximately 25 mg/Kg in accordance with the Brazilian National Malaria Control guidelines. Primaquine will be given for 7 or 14 days under supervision or not, depending on the study group. Clinical and parasitologic parameters will be monitored over a 28-day follow-up period to evaluate drug efficacy and for a total period of 168 days (24 weeks) to evaluate chances of recrudescence, relapse, or reinfection. Blood samples will be taken to measure the CQ levels in blood on Day 7 and day of failure, if occurring in the initial 28 days of follow up. In addition, a blood sample will be collected on filter paper on first day and on day of suspected failure to help differentiate parasite genotypes using techniques based on polymerase chain reaction. Results from this drug efficacy study will be used to assist the Brazilian Ministry of Health in assessing their national malaria treatment policy for P. vivax malaria.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥5 years 2. Body weight <120 kg 3. Documented fever (axillary temperature ≥37.5o C) or history of fever during the previous 48 hours in the absence of another obvious cause of fever, such as pneumonia, otitis media, etc 4. Monoinfection with P. vivax with parasitemia between 100 and 200,000 asexual parasites/µl as determined by microscopic examination of thick and thin peripheral blood smears 5. Informed consent from the patient or parent/guardian (for those <18 years), assent from child (ages 7 to 17 years inclusive), patients 5 through 6 years old will not need an assent 6. Willingness on the part of the patient to return to the clinic and/or receive home visits for regular check-ups during the 24-week (168 days) follow-up period 7. Place of residence within 30-45 minutes of study site.

Exclusion Criteria:

* 1. Presence of malaria danger signs

  1. Unable to drink
  2. Vomiting (more than twice in the previous 24 hours)
  3. Recent history of convulsions (one or more in the previous 24 hours)
  4. Impaired consciousness
  5. Unable to sit or stand 2. Presence of signs of severe malaria (WHO criteria)

  <!-- -->

  1. Cerebral malaria (unarousable coma)
  2. Severe anemia (hematocrit <15% or clinical signs) hemoglobin <5 mg/ml) (Note: we will use hemoglobin less than 8 mg/ml as exclusion criteria)
  3. Renal failure (serum creatinine >3 mg/dL or clinical signs)
  4. Pulmonary edema
  5. Hypoglycemia (blood glucose <40mg/dL or clinical signs)
  6. Shock (systolic blood pressure <70 mm Hg in adults; 50 mm Hg in children)
  7. Spontaneous bleeding/disseminate intravascular coagulation
  8. Repeated generalized convulsions
  9. Acidemia/acidosis (clinical signs)
  10. Macroscopic hemoglobinuria
  11. Jaundice 3. Self-reported presence of other underlying chronic or severe diseases (e.g., cardiac, renal, hepatic diseases, HIV/AIDS, tuberculosis, malnutrition, psoriasis) 4. History of hypersensitivity reactions to any of the drugs being tested. Mild itching with CQ is not in itself a criterion for exclusion. This occurrence will be evaluated by the study doctor before excluding the patient for this reason alone.

      5. Use of drugs with antimalarial activity in the past 30 days. (Annex D) 6. Current pregnancy (either self-reported being pregnant at enrollment or a positive urine or plasma pregnancy test at time of enrollment), previous pregnancy is not an exclusion criteria 7. Hemoglobin <8 mg/mL 8. G6PD deficiency. This will be a late exclusion criteria as soon as the results of G6PD testing becomes available.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Macedo de Oliveira, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Hospital do Jurua, Cruzeiro do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not such a plan.

REFERENCES:
- [Derived] Chamma-Siqueira NN, Negreiros SC, Ballard SB, Farias S, Silva SP, Chenet SM, Santos EJM, Pereira de Sena LW, Povoa da Costa F, Cardoso-Mello AGN, Marchesini PB, Peterka CRL, Viana GMR, Macedo de Oliveira A. Higher-Dose Primaquine to Prevent Relapse of Plasmodium vivax Malaria. N Engl J Med. 2022 Mar 31;386(13):1244-1253. doi: 10.1056/NEJMoa2104226. PMID 35353962

RESULTS

PARTICIPANT FLOW:
Groups:
- Primaquine Regular Dose Unsupervised: This is the regular primaquine dose (3.5 mg/kg) Brazil without directly observed therapy.
  Primaquine: Different total dose and supervision.
- Primaquine Regular Dose Supervised: This is the regular primaquine dose (3.5 mg/kg) in Brazil but with directly observed therapy.
  Primaquine: Different total dose and supervision.
- Primaquine Double Dose Unsupervised: This is the double total primaquine dose (14 days) (7.0 mg/kg) in Brazil with directly observed therapy.
  Primaquine: Different total dose and supervision.
Period: Overall Study
Arm/Group | Primaquine Regular Dose Unsupervised | Primaquine Regular Dose Supervised | Primaquine Double Dose Unsupervised
Started (The number of total patients included in the study (254) is different from the study because, upon review of patient records, some patients had to be excluded because they had not met the inclusion criteria.) | 63 | 96 | 95
Completed (Patient enrollment ended in October 2018, follow up ended in March 2019.) | 53 | 78 | 79
Not Completed | 10 | 18 | 16

BASELINE CHARACTERISTICS:
Population: Population of patients with vivax malaria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primaquine Regular Dose Unsupervised | Primaquine Regular Dose Supervised | Primaquine Double Dose Unsupervised | Total
Number analyzed (Participants) | 63 | 96 | 95 | 254
Age, Continuous [Median (Full Range); unit: years] | 26.5 [8.1 to 79.8] | 20.3 [5.6 to 73.9] | 23.5 [5.4 to 64.8] | 22.4 [5.4 to 79.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 44 | 43 | 115
  Male | 35 | 52 | 52 | 139
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 63 | 96 | 95 | 254

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adequate Clinical and Parasitologic Response Among Patients Enrolled
Description: Participants with adequate clinical and parasitologic response among patients enrolled, meaning patients who did not fail treatment by day 28. Those are participants who at day 28 did not present clinical deterioration or presence of parasitemia.
Time Frame: 28 days
Population: Per-protocol uncorrected analysis.
Measure: Number; unit: participants
Arm/Group | Primaquine Regular Dose Unsupervised | Primaquine Regular Dose Supervised | Primaquine Double Dose Unsupervised
Number analyzed (Participants) | 63 | 89 | 90
participants | 61 | 88 | 90

2. Primary Outcome: Participants With Adequate Clinical and Parasitologic Response Among Patients Enrolled
Description: Participants with adequate clinical and parasitologic response among patients enrolled, meaning patients who did not fail treatment by day 168. Those are participants who at day 168 did not present clinical deterioration or presence of parasitemia.
Time Frame: 168 days
Population: Per-protocol uncorrected analysis.
Measure: Number; unit: participants
Arm/Group | Primaquine Regular Dose Unsupervised | Primaquine Regular Dose Supervised | Primaquine Double Dose Unsupervised
Number analyzed (Participants) | 53 | 78 | 79
participants | 29 | 44 | 67

3. Secondary Outcome: Participants With Adequate Clinical and Parasitologic Response Based on Microsatellite-corrected Analysis Per Protocol Day 168
Description: Participants with microsatellite-corrected adequate clinical and parasitologic response among patients enrolled, meaning patients who did not fail treatment by day 168. Those are participants who at day 168 did not present clinical deterioration or presence of parasitemia with homologous (same genotype) parasites.
Time Frame: 168 days
Population: Microsatellite-corrected analysis excludes participants who, during follow-up, presented with heterologous infections (genotype different) or whose genotype could not be determined. This reduced the number of overall participants by 12 for the 'Primaquine Regular Dose Unsupervised' arm; 17 participants in the 'Primaquine Regular Dose Supervised' arm; and 8 participants in the 'Primaquine Double Dose Unsupervised' arm, in comparison to the totals in the Participant Flow section.
Measure: Number; unit: Participants
Arm/Group | Primaquine Regular Dose Unsupervised | Primaquine Regular Dose Supervised | Primaquine Double Dose Unsupervised
Number analyzed (Participants) | 41 | 61 | 71
Participants | 29 | 44 | 67

ADVERSE EVENTS:
Time Frame: During patient follow-up, 6 months.
Arm/Group | Primaquine Regular Dose Unsupervised | Primaquine Regular Dose Supervised | Primaquine Double Dose Unsupervised
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/96 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/96 | 0/95
Other Adverse Events (participants affected / at risk) | 0/63 | 0/96 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03610399/Prot_SAP_ICF_000.pdf